CLINICAL TRIAL: NCT02860026
Title: Growth and Tolerance of Healthy Term Infants Fed Cow's Milk-Based Infant Formulas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Raw ingredient shortage. Future study start date - TBD
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3388-1
Record Dates: First submitted 2016-08-03; First posted 2016-08-09 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Marketed cow's milk-based infant formula
  Interventions: Other: Marketed cow's milk-based infant formula
- Investigational (Experimental): Cow's milk-based infant formula with added nutrients
  Interventions: Other: Cow's milk-based infant formula with added nutrients

INTERVENTIONS:
Other: Marketed cow's milk-based infant formula
  Arms: Control
Other: Cow's milk-based infant formula with added nutrients
  Arms: Investigational

SUMMARY:
This clinical trial will compare the growth and tolerance of infants who consume an investigational cow's milk-based infant formula to those who consume a marketed cow's milk-based infant formula through approximately 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Singleton 10-14 days of age at randomization
* Term infant with birth weight of minimum of 2500 grams
* Solely formula fed
* Signed informed consent and protected health information

Exclusion Criteria:

* History of underlying metabolic or chronic disease, anemia, or immune compromise
* Feeding difficulties or formula intolerance

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Rate of body weight gain from 14 to 120 days of age | 3.5 months

SECONDARY OUTCOMES:
Recall of infant formula at each study visit | Up to 3.5 months
Body length measured at each study visit | Up to 3.5 months
Recall of stool characteristics questionnaire measured at each study visit | Up to 3.5 months
Head circumference measured at each study visit | Up to 3.5 months
Recall of gastrointestinal tolerance questionnaire at each study visit | Up to 3.5 months
Medically confirmed adverse events collected throughout the study period | Up to 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wu, Study Director — Mead Johnson Nutrition
Locations (17):
- United States (17):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - Altamonte Pediatric Associates, Lake Mary, Florida
  - Deaconess Clinical Research, Evansville, Indiana
  - Kentucky Pediatrics/Adult Research, Bardstown, Kentucky
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Pediatric Associates of Mt. Carmel, Inc., Cincinnati, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - UHMP Comprehensive Pediatrics, Westlake, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - The Jackson Clinic - North Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - DCOL Center for Clinical Research, Longview, Texas

IPD SHARING:
Plan to Share IPD: No